CLINICAL TRIAL: NCT01886209
Title: An Open-Label, Phase 1 Study to Examine the Pharmacokinetic Interactions Between VX-509 and Prednisone or Methylprednisolone in Healthy Male Subjects
Brief Title: Phase 1 PK Interaction Study Between VX-509 and Prednisone or Methylprednisolone in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX13-509-010
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Drug Interactions
MeSH Terms: interventions — Prednisone; 2-((2-(1H-pyrrolo(2,3-b)pyridin-3-yl)pyrimidin-4-yl)amino)-2-methyl-N-(2,2,2-trifluoroethyl)butanamide; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Prednisone 10 mg tablet on Day 1 and 7; VX-509 200 mg tablets on Days 2 thru 7
  Interventions: Drug: Prednisone; Drug: VX-509
- Cohort 2 (Experimental): Methylprednisolone 8 mg tablet on Day 1 and 7; VX-509 200 mg tablets on Days 2 thru 7
  Interventions: Drug: VX-509; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Prednisone
  Arms: Cohort 1
Drug: VX-509
Drug: Methylprednisolone
  Arms: Cohort 2

SUMMARY:
This study is designed to evaluate the effect of VX-509 on the pharmacokinetics (PK) of corticosteroids (prednisone or methylprednisolone) and the effect of corticosteroids on the PK of VX-509 and its metabolite. The study will also evaluate the safety and tolerability of VX-509 when coadministered with each of these corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18 and 55 years of age, inclusive
* Body mass index (BMI) of 18.0 to 31.0 kg/m2, inclusive, and a total body weight >50 kg

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject. This may include, but is not limited to, history of cardiovascular or central nervous system disease, diabetes, history or presence of clinically significant pathology, or history of mental disease
* Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study drug
* Subject has a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last dose of study drug
* Positive test result for any of the following infectious disease tests at the Screening Visit: T-SPOT tuberculosis (TB) test, hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus 1 and 2 antibodies

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
PK parameters including Cmax, area under the concentration-time curve from the time of dosing extrapolated to infinity (AUC0 ∞), and AUC0-last for prednisone and its metabolite prednisolone with or without VX-509 | Multiple blood samples will be obtained over the 10 day open-label treatment phase
PK parameters including Cmax, area under the concentration-time curve from the time of dosing extrapolated to infinity (AUC0 ∞), and AUC0-last for methylprednisolone with or without VX-509 | Multiple blood samples will be obtained over the 10 day open-label treatment phase

SECONDARY OUTCOMES:
Treatment-emergent adverse events, results of clinical laboratory tests, vital signs, and 12-lead electrocardiograms | Up to 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- Vertex Investigational Site, Lenexa, Kansas, United States